CLINICAL TRIAL: NCT03789955
Title: Comparison of Contralateral Oblique View With the Lateral View for Mid-thoracic Epidural Assess: a Pilot Study
Brief Title: The Superiority of Contralateral Oblique View for Mid-thoracic Epidural Assess
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Soo Choi, MD, PhD, Assistant Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-1551
Record Dates: First submitted 2018-12-27; First posted 2018-12-31 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Herpes Zoster; Postherpetic Neuralgia; Cancer
Keywords: Fluoroscopy; Contralateral Oblique View; Thoracic epidural block; Mid thoracic epidural space
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic; Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluoroscopic-guided TEB (Experimental): After assessment of the epidural space using the loss of resistance technique with air under fluoroscopic guidance, six fluoroscopic views will be obtained: true anteroposterior, contralateral oblique (CLO) at 40 degrees, 50 degrees, 60 degrees, CLO measured, and lateral for comparison CLO view with lateral view.
  Interventions: Procedure: Fluoroscopic-guided TEB

INTERVENTIONS:
Procedure: Fluoroscopic-guided TEB — When performing a fluoroscopic-guided thoracic epidural block (TEB), an 18-gauge Tuohy needle will be used for interlaminar epidural access. If the epidural space was accessed under fluoroscopic guidance and using the loss of resistance technique with air. All procedures will be performed with a paramedian approach under the true AP and lateral view at first, If the interlaminar space is not visible, the CLO view will be used. If the needle is deemed to be in the epidural space when the loss occurred, six fluoroscopic views will be obtained: true AP, CLO at 40 degrees, 50 degrees, 60 degrees, CLO measured, and lateral. The CLO measured angle will be determined by measuring the angle between the superior lamina and spinous process on the midsagittal plane on thoracic MRI or CT.

SUMMARY:
The aim of the present study is to compare contralateral oblique view with the lateral view for fluoroscopic guided mid-thoracic epidural assess.

DETAILED DESCRIPTION:
A thoracic epidural assess (block or catheter insertion) is a widely used intervention to reduce pain in patients with postherpetic neuralgia or who underwent chest and upper abdominal surgery.

In order to achieve the correct procedure, accurate access to the thoracic epidural space is needed. However, a thoracic epidural assess is a relatively more difficult procedure than procedures used in other regions, because the spinous process of the thoracic vertebra is longer than that of the lumbar vertebra, and the area through which the needle can approach the epidural space is relatively smaller due to an acute angle and larger distance between the skin and the epidural space. The midthoracic region (T4-8) is the most difficult area when performing this procedure.

To overcome this issue, a method of approaching the thoracic epidural space through the contralateral oblique view (CLO view) has been introduced, however, unlike the cervical or lumbar spine, advantages of the CLO view over the lateral view or the optimal angle of the CLO view have not yet been studied. Therefore, we planned this study to investigate the advantages of the CLO view compared with the lateral view and to determine the optimal angles of the CLO view when fluoroscopic guided mid-thoracic epidural assess.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for mid thoracic (T4-T8) epidural block or catheter insertion
* 20 ≤ age <80
* Presence of thoracic MRI or CT
* When obtaining informed consent voluntarily

Exclusion Criteria:

* Allergy to local anesthetics and contrast dye, and steroid
* Use of anticoagulants or antiplatelet medication, coagulopathy
* Infection at the insertion site
* Neurological or psychiatric disorders
* Prior spine instrumentation
* Pregnancy

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Distance between the tip of epidural needle and the baseline (CLO view - ventral interlaminar line, lateral view - spinolaminar line) at each view (CLO view at 40 degrees, 50 degrees, 60 degrees, CLO measured view, and lateral view) | One day after the procedure
  Location of the needle tip was defined as being significantly before the baseline (-2), just before the baseline (-1), on the baseline (0), just after the baseline (+1), or significantly after the baseline (+2).

SECONDARY OUTCOMES:
The quality of needle tip visualization at each view (CLO view at 40 degrees, 50 degrees, 60 degrees, CLO measured view, and lateral view) | One day after the procedure
  The clarity of the needle tip was subjectively graded as 1 (clearly visualized without ambiguity), 2 (poorly visualized or visualized with effort), or 3 (not visualized).

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Soo Choi, MD, PhD, Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan medical center, Seoul
  - Seong-Soo Choi, Seoul

REFERENCES:
- [Derived] Kim DH, Yoon SH, Lee J, Park H, Sim JH, Choi SS. Evaluation of Contralateral Oblique and Lateral Views for Mid-Thoracic Epidural Access: A Prospective Observational Study. Pain Physician. 2021 Jan;24(1):E51-E59. PMID 33400438